CLINICAL TRIAL: NCT03292393
Title: Social Norms and Antihypertensive Medication Adherence
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough sample list at participating healthcare facility.
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Health Services Research
Other Study IDs: IRB-15-0196
Record Dates: First submitted 2017-02-13; First posted 2017-09-25 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Hypertension; Medication Adherence
Keywords: Hypertension; Medication; Adherence
MeSH Terms: conditions — Hypertension; Medication Adherence | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group Contingency Management (Active Comparator): During the intervention phase, the Group Contingency Management (GCM) arm will continue to take their hypertensive medication for the four-month period and will receive a randomized phone call once a month to obtain a pill count and a home blood pressure monitoring reading using the HBPM. Participants in the GCM arm will receive a payment after each phone call, dependent on their medication adherence assessment. The GCM arm will also receive an additional payment based on their group's medication adherence.The intervention administered is the Financial Reward and Social Norms.
  Interventions: Behavioral: Financial reward; Behavioral: Social norms; Device: Home Blood Pressure Monitoring; Device: Medication adherence assessment
- Individual Contingency Management (Active Comparator): During the intervention phase, those in the Individual Contingency Management (ICM) arm will also continue to take their hypertensive medication for the four-month period but will receive a payment after each phone call, dependent on their medication adherence assessment.The intervention administered is the Financial Reward.
  Interventions: Behavioral: Financial reward; Device: Home Blood Pressure Monitoring; Device: Medication adherence assessment
- Control Arm (Placebo Comparator): During the intervention phase, those in the control arm will be asked to continue to take their hypertensive medication for the four-month period and will receive a randomized phone call once a month to obtain a pill count and a blood pressure reading using the HBPM. Those in the control arm will only be paid for their participation in the study regardless of medication adherence assessment.
  Interventions: Device: Home Blood Pressure Monitoring; Device: Medication adherence assessment

INTERVENTIONS:
Behavioral: Financial reward — In contingency management, financial rewards are contingent upon an individual changing behavior. In our study, financial incentives are contingent upon group behavioral changes.. In the intervention phase participants will be randomly assigned to one of the three treatment arms and they will receive the financial incentive that corresponds to their treatment arm. Data will be collected for four months and all participants will continue receiving a compensation for participation
  Arms: Group Contingency Management; Individual Contingency Management
Behavioral: Social norms — To build social norms the study adds a group component to a contingency management model. In contingency management, financial rewards are contingent upon an individual changing behavior. Social norms are expected to emerge as a result of the designed group contingency management, monthly-facilitated meetings at a local clinic, and daily basis interaction through social media. The intervention will build social norms that improve medication adherence of each member of a group. A three-arm randomize trial is designed to test this hypothesis. Hypertensive patients will be randomly assigned to a group contingency management (GCM) arm, an individual contingency management (ICG) arm, or a control arm.
  Arms: Group Contingency Management
Device: Home Blood Pressure Monitoring — Participants will be reminded that they will receive and learn how to use a Home Blood Pressure Monitor (HBPM) device that participant will keep for the duration of the study
Device: Medication adherence assessment — Participants will be informed that they will receive and learn how to use eCap, a medication event monitoring system that participants will return after completing the study. The project nursing student will count the number of pills the participant currently has and make a record of it on the Data Collection form.The participant will provide the project nursing student with his/her antihypertension prescription records so that the dosage amount and number of pills can be recorded on the Data Collection form.
  Other Names: eCap

SUMMARY:
The study objective is to build group social norms to improve individual adhere to antihypertensive medications. Financial incentives are provided to individuals contingent upon group behavioral changes. Groups of patients will be formed, and incentivized to interact on a daily basis through social media and participate in a monthly-facilitated meeting at a local clinic. By forming groups, making individual outcomes transparent, and setting financial incentives contingent to group targets, individual decisions are framed within emerging social norms.

DETAILED DESCRIPTION:
We propose a pilot study that will inform, provide inputs and reduce the risk of a larger implementation. The project consists of three phases: The pre-intervention phase, the intervention phase, and the post-intervention phase. The pre-intervention phase includes the recruitment and selection of participants, and a one-month collection of baseline blood pressure and medication adherence levels of participants before they are assigned to a treatment arm. All participants will receive compensation for participation.

In the intervention phase participants will be randomly assigned to one of the three treatment arms and they will receive the financial incentive that corresponds to their treatment arm. Data will be collected for four months and all participants will continue receiving a compensation for participation.

During the post-intervention phase, contingency payments will be cut off, and only compensation for participation will remain. Data will be collected for three months in the post-intervention phase.

The primary outcome of the study is medication adherence which will be measured using two different methods. The first method is through the use of eCaps (electronic caps). The second method is through a monthly randomized phone call during which the participant will be asked to perform a pill count of their medication.

The secondary outcome of the study is blood pressure which will be measured using two different instruments . The first instrument will be the ambulatory blood pressure monitor (ABPM). The second instrument will be a home blood pressure monitor (HBPM) which researchers will provide to the participant to use for the duration of the study.

All participants of the study will receive an unconditional payment each time they provide a blood pressure reading from the ABPM. Financial incentives (contingent to change in behavior -conditional to change in adherence). In addition to the unconditional payment, participants in the ICM and GCM treatment arms will receive a financial incentive that is conditional to medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Person has been diagnosed with essential hypertension for at least a year (no new or recently diagnosed hypertensive patients)
* Person is currently taking no more than 2 medications
* Person has taken the same anti-hypertensive medication for at least a year (no recent changes in medication)
* Person reports not being adherent to anti-hypertensive medication
* Speaks English or Spanish, currently insured
* Has access to the Internet
* Willing to participate in social media, able to go to West Kendall Baptist Hospital
* Available for the next 8 months

Exclusion Criteria:

* Persons with Secondary hypertension
* Persons with coronary heart disease, cerebrovascular disorders or atrial fibrillation,
* Persons with rubber allergy, or bedridden, wheelchair bound.
* Persons who have had a stroke or myocardial infarction within the previous 6 months, are pregnant, or have any serious chronic disease will also be excluded from the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Self Assessed Medication Adherence | Monthly over 8 months
  Use self reported personal pill count to calculate the Medication Possession Ratio score, this ratio is explained in the protocol and can explain how multiple measurements will be aggregated to arrive at one reported value.

SECONDARY OUTCOMES:
Self Assessed Diastolic Blood pressure (mm Hg) | Monthly over 8 months
  Self blood diastolic pressure reading with the HBPM device.
Automatic measure of Medication Adherence | Daily over 8 months
  Use the Research Electronic Data Capture (REDCap) system to gather a pill count to calculate the Medication Possession Ratio score.
Self Assessed Systolic Blood pressure (mm Hg) | Monthly over 8 months
  Self blood systolic pressure reading with the HBPM device.
Automatic measure of Diastolic Blood pressure (mm Hg) | Three times over 8 months
  Blood Diastolic pressure reading with the ABPM device.
Automatic measure of Systolic Blood pressure (mm Hg) | Three times over 8 months
  Blood Systolic pressure reading with the ABPM device.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Arrieta, PhD, Principal Investigator — Florida International University

IPD SHARING:
Plan to Share IPD: No